CLINICAL TRIAL: NCT03131063
Title: A Pilot Pharmacokinetic Study of Antibiotics in Patients Assisted by Extracorporeal Membrane Oxygenation in Intensive Care Unit
Brief Title: Pharmacokinetic Study of Antibiotics in Patients Assisted by Extracorporeal Membrane Oxygenation (PHARMECMO)
Acronym: PHARMECMO
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Responsible Party: Principal Investigator, Joe Elie Salem, MD, PhD, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: ID RCB : 2014-A00043-44
Record Dates: First submitted 2017-04-21; First posted 2017-04-27 (Actual); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Extracorporeal Membrane Oxygenation; Sepsis; Intensive Care Unit; Antibiotics
Keywords: Extracorporeal Membrane Oxygenation; Sepsis; Antibiotics; Pharmacokinetic; Intensive Care Unit
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Septic patient under ECMO treatment: Every adult patient admitted to ICU, under ECMO treatment, with known or suspected sepsis and receiving antibiotic therapy, was eligible for inclusion. The concentration of the studied antibiotics was determined by a combination of liquid chromatography and mass spectrometry from blood samples. For intermittent administration of antibiotic, two successive samples were performed both at 50% (Cmax) and 100% (Cmin) of the dosing interval.
  Interventions: Other: Antibiotic plasma dosage

INTERVENTIONS:
Other: Antibiotic plasma dosage — Measurement of the concentration of antibiotics administered as part of the routine care of intensive care patients

SUMMARY:
The PHARMECMO study is a pilot, prospective, pharmacokinetic study, conducted in a cardiac surgery intensive care unit of 18 beds. Optimization of antibiotic therapy for extracorporeal membrane oxygenation (ECMO) patients remains a pharmacological challenge. Clinical studies suggest that individualized dosing strategies and therapeutic drug monitoring could facilitate the achievement of adequate antibiotic concentration. The objective of this pilot study was to observe the pharmacokinetic characteristics of commonly used antibiotics in intensive care for patients treated with extracorporeal membrane oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Extra corporeal membrane oxygenation treatment
* Parenteral antibiotherapy for known or suspected sepsis
* Informed consent

Exclusion Criteria:

* Refusal of participation
* Pregnancy
* Burned patient
* Steady state conditions not reached
* Non-intravenous administration of antibiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were selected from patients hospitalized in cardiac surgical intensive care units with clinico-biological elements in favor of sepsis and for whom antibiotic therapy was instituted. An ECMO treatment before study enrollement was required.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Minimum Antibiotics plasma concentration (Cmin) (C min) | Up to 24 hours
  Dosage under steady state conditions of every antibiotics plasma concentration just before the next administration in patients with sepsis and treated by ECMO
Medium Antibiotics plasma concentration (CT 50) | Up to 24 hours
  Dosage under steady state conditions of every antibiotic plasma concentration in the middle of the interval between two administration (CT 50) in patients with sepsis and treated by ECMO

CONTACTS AND LOCATIONS:
Overall Officials: Amour Julien, MD, PhD, Study Director — Hôpital Universitaire La Pitié-Salpêtrière, Assistance Publique - Hôpitaux de Paris, Faculté de médecine, Université Pierre et Marie Curie, Paris, INSERM U1166-ICAN, France

IPD SHARING:
Plan to Share IPD: No